CLINICAL TRIAL: NCT05832515
Title: Trial of the Efficacy and Safety of High-dose Immunosuppressive Therapy Based on Fludarabine and Cyclophosphamide-containing Conditioning Regimen Followed by Autologous Hematopoietic Stem Cell Transplantation in Patients With Multiple Sclerosis.
Brief Title: AHSCT With Fludarabine and Cyclophosphamide Based Conditioning Regimes in Patients With Multiple Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FluCy_MS
Record Dates: First submitted 2022-04-04; First posted 2023-04-27 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Autoimmune Diseases; AHSCT; Fludarabine
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases | interventions — fludarabine phosphate; Injections; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AHSCT: FluCy200 (Experimental): AHSCT with reduced intensity condition regimen (RIC):
  cyclophosphamide intravenously at a dose of 50 mg/kg/day from -5 to day -2 inclusive; fludarabine intravenously at a dose of 30 mg/m2 from -5 to day -2 inclusive. Immunotherapy: ATG - ATGAM intravenously 20 mg/kg from -3 to -1 or Thymoglobulin 2.5 mg/kg from -3 to -1 day.
  Also, within the framework of immunotherapy, instead of ATG, it is allowed to use anti-B-cell therapy - Rituximab 500 mg / m2 per day +12 AHSCT.
  Interventions: Drug: Fludarabine Phosphate for Injection

INTERVENTIONS:
Drug: Fludarabine Phosphate for Injection — Intravenous injection of fludarabine phosphate at a dose of 30 mg/m2 from day -5 to day -2 of immunoablative conditioning regimen.
  Other Names: Fludarabine

SUMMARY:
One of the possible options for the treatment of MS at present is a high-dose immunosuppressive therapy followed by autologous hematopoietic stem cell transplantation (HIST-AHSCT), which is a highly effective treatment for patients with relapsing-remitting MS.

This method of MS treatment was introduced in 1997. Significant complications and mortality associated with HIST-ATHSC is an obstacle to broad use of this method. The risk is even greater in patients with advanced disease, long duration of previous treatment and aggressive forms of MS.

Despite toxicity certain progressive cases of MS are still an indication for HIST-autoHSCT.

Most commonly used conditioning regimens for multiple sclerosis include high-dose cyclophosphamide. One of the options to reduce cyclophosphamide-related toxicity and dose is addition of fludarabine. Fludarabine is a cytostatic drug, an antimetabolite from the group of purine antagonists. It has a pronounced immunosuppressive activity and no overlapping toxicity with cyclophosphamide. The study will evaluate the safety and efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65;
* 1.0-6.5 points on the EDSS scale (for MS);
* Length of illness - any;
* Disease progression during the last 6 months while taking drugs of 1st and 2nd lines;
* An established and confirmed diagnosis of an autoimmune disease in the previous stages of treatment;
* Ineffectiveness, inaccessibility or intolerance of Disease-Modifying Therapies;
* Relapse after AHSCT.
* Absence of severe concomitant somatic pathology;
* Left ventricular injection fraction > 50%;
* Karnofsky Performance Score (KPS) > 30%;
* The ability to take oral medications;
* Life expectancy is more than 1 month;
* Signed informed consent of the patient or legal representatives.

Exclusion Criteria:

* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky performans status <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Multiple sclerosis progression free survival | 365 days
  To evaluate safety and effectiveness of immunoablative conditioning regimen FluCy200 in patients with refractory multiple sclerosis after AHSCT.

SECONDARY OUTCOMES:
Cumulative incidence of mortality | 365 days
  Death from any cause after AHSCT
To evaluate adverse effects after FluCy200 conditioning regimen | 365 days
  Toxicity based NCI CTCAE ver.5.0, including analysis of severe bacterial, fungal and viral infections incidence
Quality of life status 1 | 365 days
  Multiple sclerosis-specific questionnaire - HADS (Hospital Anxiety and Depression Scale) before and after AHSCT:
  0-7 points - normal; 8-10 - subclinically expressed anxiety/depression; 11-21 - clinically expressed anxiety/depression.
Quality of life status 2 | 365 days
  Multiple sclerosis-specific questionnaire - The Short Form-36 (SF-36) before and after AHSCT: The SF-36 consists of 36 questions grouped into eight scales: physical functioning, role-physical functioning, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The indicators of each scale are compiled in such a way that the higher the value of the indicator (from 0 to 100), the better the score on the chosen scale. Of these, two parameters are formed: the psychological and physical components of health.
Quality of life status 3 | 365 days
  Multiple sclerosis-specific questionnaire - Multiple Sclerosis Impact Scale (MSIS-29) before and after AHSCT:
  The MSIS-29 scale consists of 29 items and includes indicators observed over the previous two weeks, including 20 of which characterize physical condition, coordination and mobility, and 9 questions reflect the patient's mental state. Answers are ranked on a 5-point Likert scale from 1 to 5 (1 = none; 2 = little; 3 = moderate; 4 = significant; 5 = very strong) in one direction.
  The total score is the sum of all 29 responses and can range from 29 to 145. A higher score means a higher degree of disability. The result is assessed on a scale from 0 to 100, where a higher result means worse health.
Quality of life status 4 | 365 days
  Multiple sclerosis-specific questionnaire - Functional Assessment of Multiple Sclerosis (FAMS) before and after AHSCT:
  FAMS Total score (range=0-176) is derived by adding: 1) Mobility (r=0-28). 2) Symptoms (r=0-28). 3) Emotional well- being (r=0-28). 4) General contentment (r=0-28). 5) Thinking and fatigue (r=0-36). 6) Family/social wellbeing (r=0-28).
  Higher scores indicate better quality of life.
Neurological status 1 | 365 days
  Multiple sclerosis-specific questionnaire - EDSS (Expanded Disability Status Scale) before and after AHSCT:
  0 points - Normal neurologic exam; 1.0-1.5 - No disability, minimal signs in one or two Functional Systems (FS); 2.0-2.5 - Minimal disability in one or two FS; 3.0-3,5 - Moderate disability in one FS, fully ambulatory; 4.0-4.5 - Fully ambulatory without aid. Able to walk without aid or rest some 500 or 300 meters; 5.0-5.5 - Ambulatory without aid or rest for about 200 or 100 meters; 6.0 - Intermittent assistance required to walk about 100 meters; 6.5 - Constant bilateral assistance required to walk about 20 meters; 7.0-7.5 - Unable to walk beyond about 5 meters or more than a few steps; 8.0 - Essentially restricted to bed, but may be out of bed itself; 8.5 - Essentially restricted to bed; 9.0 - Helpless bed patient; can communicate and eat; 9.5 - Totally helpless bed patient; unable to communicate effectively or eat/swallow; 10 - Death due to MS
Immune reconstitution | 365 days
  Absolute number of CD3+, CD4+, CD8+, CD45+, CD19+ T-lymphocytes in cells/ml
Magnetic resonance imaging response | 365 days
  Measured by Magnetic Resonance Disease Severity Scale (MRDSS)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan S Moiseev, Principal Investigator — Pavlov First Saint Petersburg State Medical University
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia